CLINICAL TRIAL: NCT06543082
Title: Clinical Outcomes of Colchicine Therapy Following Percutaneous Coronary Intervention in Patients With Acute Coronary Syndrome: the MACT (Mono Antiplatelet and Colchicine Therapy) Prospective Multicenter Study
Brief Title: MACT (Mono Antiplatelet and Colchicine Therapy) Prospective Multicenter Study
Acronym: MACT II
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: CHA University (Other)
Collaborators: Biotronik SE & Co. KG (Industry)
Responsible Party: Principal Investigator, Seung-Yul Lee, Associate Professor, Division of Cardiology, Department of Internal Medicine, CHA University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHAMC IRB 2024-01-057-009
Record Dates: First submitted 2024-08-03; First posted 2024-08-07 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Acute Coronary Syndrome
Keywords: Colchicine
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Colchicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MACT (Experimental): Mono Antiplatelet and Colchicine Therapy
  Interventions: Drug: Colchicine 0.6 mg

INTERVENTIONS:
Drug: Colchicine 0.6 mg — Participants will take low-dose colchicine (0.6 mg once daily) in addition to ticagrelor maintenance therapy (90 mg twice daily), and discontinue aspirin the day after PCI. They will have an hs-CRP test 1 month after PCI. If the hs-CRP level is below 2 mg/L, colchicine will be discontinued 1 month after PCI. If it is 2 mg/L or higher, colchicine will be continued for 12 months after PCI.

SUMMARY:
The previous Mono Antiplatelet and Colchicine Therapy (MACT) pilot study (NCT04949516) demonstrated that it was feasible to discontinue aspirin therapy and administer low-dose colchicine on the day after percutaneous coronary intervention (PCI) in addition to potent P2Y12 inhibitors in patients with acute coronary syndrome (ACS). However, the efficacy and safety of MACT have not yet been investigated. The goal of this clinical trial is to evaluate the clinical outcomes of ticagrelor P2Y12 inhibitor monotherapy combined with colchicine immediately after PCI in patients with ACS. The main questions it aims to answer are:

* What is the frequency of the composite endpoint of cardiovascular death, nonfatal spontaneous myocardial infarction, nonfatal ischemic stroke, unplanned hospitalization leading to urgent revascularization, and major bleeding at 12 months post-intervention?
* What is the frequency of stent thrombosis at 12 months post-intervention?

For pre-specified analyses, researchers will compare MACT to less than 1 month, 3-month, and 12-month dual antiplatelet therapy (individual patient data from the T-PASS [NCT03797651] and TICO [NCT02494895] trials) to determine if MACT is effective in treating ACS.

Participants will:

* Take low-dose colchicine in addition to ticagrelor maintenance therapy, discontinuing aspirin the day after PCI.
* Take a high-sensitivity C-reactive protein (hs-CRP) test 1 month after PCI.
* Discontinue colchicine if the hs-CRP level is less than 2 mg/L, or continue colchicine if it is not.
* Visit the clinic for check-ups at 1, 3, 6, 9, and 12 months after PCI.

ELIGIBILITY:
Inclusion Criteria:

* Participants with positive troponin acute coronary syndrome who have undergone implantation of ultrathin bioresorbable polymer sirolimus-eluting stents (Orsiro; Biotronik AG).
* Participants who have provided written informed consent.

Exclusion Criteria:

* Under 19 years of age.
* Stent treatment failure lesions (stent restenosis or thrombosis).
* Cardiac arrest or cardiogenic shock.
* Currently taking or requiring strong CYP3A4 inhibitors (atazanavir, clarithromycin, darunavir/ritonavir, indinavir, itraconazole, ketoconazole, lopinavir/ritonavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, tipranavir/ritonavir) or P-glycoprotein inhibitors (cyclosporine, ranolazine).
* Presence of any of the following concomitant conditions: myelosuppression, leukopenia, granulocytopenia, thrombocytopenia, pancytopenia, aplastic anemia, severe gastrointestinal diseases, or genetic disorders such as galactose intolerance.
* Hypersensitivity to colchicine treatment.
* Currently taking colchicine for another condition.
* Requiring anticoagulant therapy.
* Liver disease classified as Child-Pugh class B or C.
* Renal disease with creatinine clearance <50 mL/min.
* Pregnant, breastfeeding, or women of childbearing age.
* Currently has a malignancy or has a history of malignancy within the past 5 years.
* Life expectancy of less than 5 years.
* Contraindication for ticagrelor use (history of intracranial hemorrhage, active pathological bleeding, or liver disease classified as Child-Pugh class B or C).

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy Outcome: Net adverse clinical event | 12 months post-intervention
  The composite of cardiovascular death, nonfatal spontaneous (nonprocedural) myocardial infarction, nonfatal ischemic stroke, unplanned hospitalization leading to urgent revascularization, and major bleeding
Safety Outcome: Stent thrombosis | 12 months post-intervention
  Definite, probable, or possible stent thrombosis according to the Academic Research Consortium

SECONDARY OUTCOMES:
Cardiovascular death | 12 months post-intervention
  The composite of cardiac and vascular death. Any death due to proximate cardiac cause (eg, myocardial infarction, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, and all procedure-related deaths, including those related to concomitant treatment, will be classified as cardiac death. Death caused by noncoronary vascular causes, such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular diseases will be classified as vascular death.
Nonfatal spontaneous (nonprocedural) myocardial infarction | 12 months post-intervention
  Myocardial infarction is defined as symptoms, electrocardiographic changes, or abnormal imaging findings, combined with a creatine kinase MB fraction above the upper normal limits or a troponin T or troponin I level greater than the 99th percentile of the upper normal limit. Myocardial infarction that are not associated with a revascularization procedure will be classified as nonfatal spontaneous myocardial infarction.
Nonfatal ischemic stroke | 12 months post-intervention
  Cerebrovascular event resulting in a neurologic deficit within 24 hours or the presence of acute infarction as demonstrated by imaging studies will be classified as nonfatal ischemic stroke.
Unplanned hospitalization leading to urgent revascularization | 12 months post-intervention
  This event will be present only if the participant is hospitalized unexpectedly because of persisting or increasing complaints of chest pain (with or without ST-T changes, with or without elevated biomarkers) and a revascularization is performed within the same hospitalization. It should be clearly distinguished from the revascularization procedure which is performed on non-urgent basis.
Major bleeding | 12 months post-intervention
  Bleeding Academic Research Consortium type 3 or 5
High residual inflammation | 1 month, 6 months, and 12 months post-intervention
  Participant with hs-CRP of ≥2 mg/L
High residual platelet reactivity | 1 month and 12 months post-intervention
  Participant with P2Y12 reaction units of >208
Low residual platelet reactivity | 1 month and 12 months post-intervention
  Participant with P2Y12 reaction units of <85
Thrombogenicity | 1 month and 12 months post-intervention
  This will be measured using R, K, Angle, A10, MA, and Ly30 through thromboelastography.
Adverse drug reaction to colchicine | 1 month, 3 months, 6 months, 9 months, and 12 months
  Response to a colchicine which is noxious and unintended and which occurs during the administration period.

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Yul Lee, MD, Principal Investigator — CHA Bundang Medical Center
Locations (1):
- CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee SY, Jeong YH, Yun KH, Cho JY, Gorog DA, Angiolillo DJ, Kim JW, Jang Y. P2Y12 Inhibitor Monotherapy Combined With Colchicine Following PCI in ACS Patients: The MACT Pilot Study. JACC Cardiovasc Interv. 2023 Aug 14;16(15):1845-1855. doi: 10.1016/j.jcin.2023.05.035. PMID 37587591
- [Background] Lee SY, Cho JY, Gorog DA, Angiolillo DJ, Yun KH, Ahn JH, Koh JS, Park Y, Hwang SJ, Hwang JY, Kim JW, Jang Y, Jeong YH. Inflammation and platelet reactivity during adjunctive colchicine versus aspirin in patients with acute coronary syndrome treated with potent P2Y12 inhibitor. Front Med (Lausanne). 2024 Apr 19;11:1349577. doi: 10.3389/fmed.2024.1349577. eCollection 2024. PMID 38841588
- [Background] Kim BK, Hong SJ, Cho YH, Yun KH, Kim YH, Suh Y, Cho JY, Her AY, Cho S, Jeon DW, Yoo SY, Cho DK, Hong BK, Kwon H, Ahn CM, Shin DH, Nam CM, Kim JS, Ko YG, Choi D, Hong MK, Jang Y; TICO Investigators. Effect of Ticagrelor Monotherapy vs Ticagrelor With Aspirin on Major Bleeding and Cardiovascular Events in Patients With Acute Coronary Syndrome: The TICO Randomized Clinical Trial. JAMA. 2020 Jun 16;323(23):2407-2416. doi: 10.1001/jama.2020.7580. PMID 32543684
- [Background] Hong SJ, Lee SJ, Suh Y, Yun KH, Kang TS, Shin S, Kwon SW, Lee JW, Cho DK, Park JK, Bae JW, Kang WC, Kim S, Lee YJ, Ahn CM, Kim JS, Kim BK, Ko YG, Choi D, Jang Y, Hong MK; T-PASS (Ticagrelor Monotherapy in Patients Treated With New-Generation Drug-Eluting Stents for Acute Coronary Syndrome) Investigators. Stopping Aspirin Within 1 Month After Stenting for Ticagrelor Monotherapy in Acute Coronary Syndrome: The T-PASS Randomized Noninferiority Trial. Circulation. 2024 Feb 20;149(8):562-573. doi: 10.1161/CIRCULATIONAHA.123.066943. Epub 2023 Oct 25. PMID 37878786
- [Background] Cutlip DE, Windecker S, Mehran R, Boam A, Cohen DJ, van Es GA, Steg PG, Morel MA, Mauri L, Vranckx P, McFadden E, Lansky A, Hamon M, Krucoff MW, Serruys PW; Academic Research Consortium. Clinical end points in coronary stent trials: a case for standardized definitions. Circulation. 2007 May 1;115(17):2344-51. doi: 10.1161/CIRCULATIONAHA.106.685313. PMID 17470709
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Derived] Jang JY, Suh Y, Kim C, Byoun JT, Yun KH, Lee JH, Jeon KH, Cho S, Yoon HJ, Kim JW, Lee B, Kang SH, Kim SH, Moon JY, Jang Y, Lee SY. Efficacy and safety of mono antiplatelet therapy with colchicine in acute coronary syndrome patients following percutaneous coronary intervention: rationale and design of the MACT II trial. Front Cardiovasc Med. 2025 Oct 27;12:1662392. doi: 10.3389/fcvm.2025.1662392. eCollection 2025. PMID 41221450
- See also: The MACT Pilot Study — http://pubmed.ncbi.nlm.nih.gov/37587591/